CLINICAL TRIAL: NCT03646240
Title: Phase 1 Study of ABI-009 (Nab-rapamycin) for Surgically-Refractory Epilepsy (RaSuRE)
Brief Title: ABI-009 (Nab-rapamycin) for Surgically-Refractory Epilepsy (RaSuRE)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Aadi Bioscience, Inc. (Industry)
Responsible Party: Principal Investigator, Jason Hauptman, Attending Pediatric Neurosurgeon, Seattle Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RaSuRE
Record Dates: First submitted 2018-07-19; First posted 2018-08-24 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Epilepsy Intractable
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Intervention Model Description: Participation includes a 4-week baseline period, a 3-week dosing period and a 12-week follow-up period. After baseline participants will receive ABI-009 given weekly IV for 3 weeks. ABI-009 will be tested in cohorts of 3 participants using the standard 3+3 dose-finding design.
  Escalation to the next dose level with a new cohort of 3 participants will occur after no DLT was observed. There will be no intra-participant dose escalation allowed. If DLT occurs in a cohort, an additional 3 participants will be recruited to the cohort. If no further DLTs occur, a new cohort of 3 participants at the next higher dose level can be enrolled. If 2/6 participants at dose level 1 experience a DLT, then that cohort will be closed to further enrollment and 3 participants will be enrolled at the next lower dose level, and so on. The MTD is the highest dose level in which ≤1 participant has a DLT.
  Once MTD has been determined, MTD cohort will be opened for up to 6 additional participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dosing arm (Experimental)
  Interventions: Drug: ABI-009

INTERVENTIONS:
Drug: ABI-009 — For dose finding, ABI-009 will start at 5 mg/m2/dose IV, once a week for three weeks, in cohorts of 3 participants each using the standard 3+3 dose-finding design

SUMMARY:
This is a prospective, single-center, phase 1 safety study to investigate the safety, tolerability, seizure control, and quality of life in participants with medically-refractory epilepsy who failed epilepsy surgery. These participants will have continued seizures despite being at least 3 months post-epilepsy surgery (resective surgery with an intent to cure).

DETAILED DESCRIPTION:
Seizures that are refractory to both medical and surgical therapy increase the risk of morbidity and mortality in children with epilepsy. At this point in time, options for these children are sparse and suboptimal. This hypothesis-driven phase 1 study aims to evaluate the use of a mammalian target of rapamycin [mTOR] inhibitor, ABI-009, in this subset of challenging participants. The underlying hypotheses being tested in trial are: (1) ABI-009 is a safe and well-tolerated medication in children who have medically-refractory epilepsy and have failed epilepsy surgery, and (2) The addition of ABI-009 therapy to the current clinical standard of continued antiepileptic medications results in improved epilepsy control. This is unique among trials of anti-epileptic medications in that it also studies mTOR inhibition in a non-Tuberous Sclerosis Complex (TSC) specific population for whom few additional effective therapies exist.

Upon enrollment, participants will be continued and observed on their pre-existing, clinically prescribed antiepileptic drug (AED) regimen for 1 month. At the 1-month mark, participants will receive weekly ABI-009 intravenously at different dose levels in cohorts of 3 participants each using the standard 3+3 dose-finding design. ABI-009 will be continued for a total of 3 weeks. ABI-009 will then be discontinued and the participants will be observed for an additional 3 months. The investigators intend an expansion of the maximum tolerated dose (MTD) cohort to an estimated additional 6 participants for a maximum possible enrollment of 18 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent (and assent when applicable) obtained from participant or participant's legal representative
2. Be willing and able to adhere to the study visit schedule and other protocol requirements
3. Male or female ≥3 and ≤26 years of age at Visit 1 b. Because no dosing or adverse event data are currently available on the use of ABI-009 or other mTOR inhibitors in participants <3 years of age, these young children are excluded from this study.
4. Documentation of a diagnosis of medically intractable epilepsy as defined by the failure of at least 2 appropriately dosed and tolerated AEDs to eliminate all clinical seizures over a 6-month period (prior to epilepsy surgery)
5. Documentation of resective epilepsy surgery following appropriate pre-surgical evaluation
6. Documentation of continued clinical seizures that persist at least 3 months following resective epilepsy surgery. In order to proceed with drug administration, participants will have to have had >8 seizures in the last 30 days without 2 weeks of seizure freedom, as noted by a daily seizure diary.
7. Documentation that the participant is not a candidate for OR refuses any additional resective epilepsy surgery
8. Participants must have adequate bone marrow function (ANC ≥1,000/mm3, platelet count of ≥100,000/mm3, and hemoglobin ≥9 gm/dL) before starting study drug.
9. Participants must have adequate liver function (SGPT/ALT ≤5 times ULN and bilirubin ≤5 times ULN) before starting study drug.
10. Participants must have adequate renal function, defined as: Creatinine clearance or radioisotope GFR >/= 70mL/min/1.73 m2 or a serum creatinine based on age/gender as follows:
11. Participants must have a fasting cholesterol level <350 mg/dL and triglycerides <400 mg/dL before starting study drug. In case one or both of these are exceeded, the participant can only be included after initiation of appropriate lipid lowering medication and documentation of cholesterol <350mg/dL and triglycerides <400mg/dl before start of study drug.
12. Participants must have normal oxygen saturation.
13. The effects of ABI-009 on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because rapamycin is known to be teratogenic, female participants of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a female participant become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

    1. Participants of child bearing potential must not be breastfeeding or pregnant as evidenced by a negative pregnancy test.

Exclusion Criteria:

1. For females of child bearing potential:

   1. Positive pregnancy test at Visit 1, or
   2. Lactating, or
   3. Unwilling to practice a medically acceptable form of contraception (acceptable forms of contraception: abstinence, hormonal birth control, intrauterine device, or barrier method plus a spermicidal agent), unless surgically sterilized or postmenopausal during the study.
2. Has any other condition that, in the opinion of the Site Investigator/designee, would preclude informed consent or assent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.
3. Participants should not receive immunization with attenuated live vaccines within one week of study entry or during study period. Close contact with those who have received attenuated live vaccines should be avoided during the ABI-009 dosing period. Examples of live vaccines include intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella and TY21a typhoid vaccines.
4. HBsAg and HCVAb blood test must be done at screening (HBsAg only needs to be screened in patients who have not received the full complement of Hepatitis B immunizations). Patients who test positive for Hepatitis C antibodies or the Hepatitis B antigen are ineligible. Alternatively, if the patient has received the complement of Hepatitis B immunizations, this would suffice.
5. A known history of HIV seropositivity. HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with ABI-009. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.
6. Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent. Note: Patients that are currently using inhaled, intranasal, ocular, topical or other non-oral or non-IV steroids are not necessarily excluded from the study but need to be discussed with the study chair.
7. Patients who have been previously treated with a systemic mTOR inhibitor for epilepsy. Skin cream use with rapamycin or everolimus, however, is permitted.
8. Patients with a known hypersensitivity to human albumin, ABI-009 or other rapamycins (e.g. sirolimus, everolimus, temsirolimus).
9. Patients receiving any other concurrent anticancer or investigational therapy. Participants will be permitted to enroll in the study after a 30-day washout of previously used investigational drugs.
10. Patients with any clinically significant unrelated systemic illness that would compromise a participant's ability to tolerate protocol procedures.
11. Patients with inability to return for dosing and follow-up visits to assess toxicity to the study drug.
12. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, active lung disease, or psychiatric illness/social situations that would limit compliance with study requirements. Study Specific Tolerance for Inclusion/Exclusion Criteria Patients who fail to meet one or more of the inclusion criteria or who meet any of the exclusion criteria will not be enrolled in this study. Waivers of any of the above study entry criteria will not be granted.

Ages: 3 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 3 weeks
  Incidence of AEs in each treatment arm will be tabulated by seriousness, severity, and relationship to study drug from baseline will be summarized by treatment group.

SECONDARY OUTCOMES:
Percentage reduction in seizure rate | 4 months
  Frequency measured using median percentage reduction

CONTACTS AND LOCATIONS:
Overall Officials: Jason Hauptman, MD, PhD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/40/NCT03646240/Prot_SAP_000.pdf